CLINICAL TRIAL: NCT00496262
Title: Pharmacokinetics of Haemocomplettan® P in Subjects With Congenital Fibrinogen Deficiency
Brief Title: Human Fibrinogen - Pharmacokinetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI3023_2001
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2009-07-10 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2011-02

CONDITIONS: Fibrinogen Deficiency
Keywords: Congenital fibrinogen deficiency; Fibrinogen concentrate; Pharmacokinetics; Thrombelastography
MeSH Terms: conditions — Afibrinogenemia | interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human Fibrinogen Concentrate (Experimental)
  Interventions: Biological: Human Fibrinogen Concentrate

INTERVENTIONS:
Biological: Human Fibrinogen Concentrate — Single intravenous infusion of 70 mg/kg body weight
  Other Names: Haemocomplettan® P; RiaSTAP

SUMMARY:
This study evaluated the single-dose pharmacokinetics of human fibrinogen concentrate and clot strength (maximum clot firmness [MCF]) in subjects with congenital fibrinogen deficiency. MCF was measured to demonstrate the functional activity of replacement fibrinogen when a fixed dose of human fibrinogen concentrate was administered.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 6 years
* Documented congenital fibrinogen deficiency: fibrinogen deficiency manifested as afibrinogenemia with plasma fibrinogen activity and antigen at screening undetectable (i.e. < 20 mg/dL)
* Informed consent signed by subject or legal guardian

Exclusion Criteria:

* Presence or history of hypersensitivity to Human Fibrinogen Concentrate or human plasma proteins,
* Presence or history of deep vein thrombosis, pulmonary embolism, or arterial thrombosis
* Acute bleeding
* History of esophageal varicose bleeding
* End stage liver disease (i.e. Child-Pugh score B or C)
* Planned major surgery with a need for blood transfusion during the PK blood sampling period
* Polytrauma within 1 year prior to enrollment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (15):
- United States (6):
  - Contact CSL Behring for facility details, Aurora, Colorado
  - Contact CSL Behring for facility details, St. Petersburg, Florida
  - Contact CSL Behring for facility details, Chicago, Illinois
  - Contact CSL Behring for facility details, Scarborough, Maine
  - Contact CSL Behring for facility details, New York, New York
  - Contact CSL Behring for facility details, Pittsburgh, Pennsylvania
- Italy (9):
  - Contact CSL Behring for facility details, Cagliari
  - Contact CSL Behring for facility details, Florence
  - Contact CSL Behring for facility details, Milan
  - Contact CSL Behring for facility details, Napoli
  - Contact CSL Behring for facility details, Padua
  - Contact CSL Behring for facility details, Palermo
  - Contact CSL Behring for facility details, Rome
  - Contact CSL Behring for facility details, Sassari
  - Contact CSL Behring for facility details, Vicenza

REFERENCES:
- [Result] Manco-Johnson MJ, Dimichele D, Castaman G, Fremann S, Knaub S, Kalina U, Peyvandi F, Piseddu G, Mannucci P; FIBRINOGEN CONCENTRATE STUDY GROUP. Pharmacokinetics and safety of fibrinogen concentrate. J Thromb Haemost. 2009 Dec;7(12):2064-9. doi: 10.1111/j.1538-7836.2009.03633.x. Epub 2009 Oct 5. PMID 19804533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at study sites in the USA and Italy.
Groups:
- Human Fibrinogen Concentrate: All enrolled subjects received a single IV infusion of 70 mg/kg body weight of human fibrinogen concentrate.
Period: Overall Study
Arm/Group | Human Fibrinogen Concentrate
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Human Fibrinogen Concentrate: Includes all subjects who received any portion of the infusion of human fibrinogen concentrate.
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (15.9)
Age, Customized [Number; unit: participants]
  <16 years | 4
  ≥16 to < 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Clot Firmness (MCF)
Description: MCF is a functional parameter that depends on the activation of coagulation, the fibrinogen content of the sample (in plasma), and the polymerization and crosslinking of the fibrin network. MCF was determined by rotational thromboelastometry (ROTEM) testing.
Time Frame: Pre-infusion and 1 hour post-infusion
Population: All subjects in the intention to treat (ITT) population. The ITT population included all subjects who received any portion of any infusion of human fibrinogen concentrate. (Note: 2 subjects in the ITT population had missing MCF data; the change from baseline MCF was entered as 0.0 for these subjects.)
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Pre-infusion: ≤ 2 hours before start of infusion
- 1 Hour Post-infusion: 1 hour after end of infusion
Arm/Group | Pre-infusion | 1 Hour Post-infusion
Number analyzed (Participants) | 15 | 15
millimeters | 0 (0) | 8.9 (4.4)
Statistical Analysis 1: Comparison: Pre-infusion vs 1 Hour Post-infusion; This is an open-label study with statistical comparison between MCF pre-infusion and 1 hour post-infusion; Test type: Superiority or Other; p < 0.0001, 2-sided, 1-sample t-test; Mean Difference (Net) = 8.9, Standard Deviation 4.4 — The entire ITT population was used for a conservative analysis of the mean change in MCF. The mean change was set to 0 for any subject with missing MCF data

2. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: t1/2 for fibrinogen activity was determined from samples taken at 12 timepoints during the specified time frame.
Time Frame: 0.5 hours to 13 days post-infusion
Population: The pharmacokinetic analysis population (PK PP) included all subjects who received >90% of the infusion and who also had sufficient data for a reliable PK analysis (n=14).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
hours | 78.7 (18.1)

3. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax for fibrinogen activity was determined from samples taken at 12 timepoints during the specified time frame.
Time Frame: Pre-infusion to 13 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
g/L | 1.4 (0.27)

4. Secondary Outcome: Area Under the Concentration-time Curve (AUC) Standardized for 70 mg/kg Body Weight Dose
Description: AUC for fibrinogen activity was determined from samples taken at 12 timepoints during the specified time frame.
Time Frame: Pre-infusion to 13 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*mg/mL
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
hour*mg/mL | 124.3 (24.16)

5. Secondary Outcome: Clearance (Cl)
Description: Cl for fibrinogen activity was determined from samples taken at 12 timepoints during the specified time frame.
Time Frame: Pre-infusion to 13 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/hour/kg
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
mL/hour/kg | 0.59 (0.13)

6. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT for fibrinogen activity was determined from samples taken at 12 timepoints during the specified time frame.
Time Frame: Pre-infusion to 13 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
hours | 92.8 (20.1)

7. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Vss for fibrinogen activity was determined from samples taken at 11 timepoints during the specified time frame.
Time Frame: Pre-infusion to 13 days post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
mL/kg | 52.7 (7.48)

8. Secondary Outcome: Incremental In Vivo Recovery (IVR)
Description: Maximum fibrinogen activity increase in plasma per mg/kg dosed
Time Frame: Pre-infusion to 4 hours post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL increase per mg/kg body weight
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
mg/dL increase per mg/kg body weight | 1.7 [1.3 to 2.7]

9. Secondary Outcome: Classical In Vivo Recovery (IVR)
Description: Maximum fibrinogen activity increase in plasma times plasma volume per mg/kg dose
Time Frame: Pre-infusion to 4 hours post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: % of expected increase in fibrinogen
Arm/Group | Human Fibrinogen Concentrate
Number analyzed (Participants) | 14
% of expected increase in fibrinogen | 61.8 [52.5 to 97.4]

ADVERSE EVENTS:
Arm/Group | Human Fibrinogen Concentrate
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Fibrinogen Concentrate (N=15)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned before seeking publication review.